CLINICAL TRIAL: NCT01672008
Title: A Phase IIa Study of Safety and Efficacy of NOX-100 for Preventing Hypotension in Patients During Hemodialysis Sessions
Brief Title: NOX-100 for Preventing Hypotension During Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medinox, Inc. (Industry)
Collaborators: Orient Europharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NOX-100-ORIENT201
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Hypotension
Keywords: NOX-100
MeSH Terms: conditions — Hypotension | interventions — nitric oxide scavenger 100

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NOX-100/Placebo (Experimental): After enrollment, subjects will be randomly assigned to one of the following treatment sequences in a 1:1 ratio.
  Sequence A: NOX-100 treatment phase followed by Placebo treatment phase Sequence B: Placebo treatment phase followed by NOX-100 treatment phase
  Interventions: Drug: NOX-100
- Placebo/NOX-100 (Experimental): After enrollment, subjects will be randomly assigned to one of the following treatment sequences in a 1:1 ratio.
  Sequence A: NOX-100 treatment phase followed by Placebo treatment phase Sequence B: Placebo treatment phase followed by NOX-100 treatment phase
  Interventions: Drug: NOX-100

INTERVENTIONS:
Drug: NOX-100

SUMMARY:
This study is designed to evaluate the safety, tolerability and efficacy profile of NOX-100 to reduce intradialytic hypotension (IDH) in patients undergoing chronic hemodialysis (HD).

DETAILED DESCRIPTION:
This is a 2-stage, prospective, randomized, double-blind, multi-dose, placebo-controlled, cross-over, phase IIa study to evaluate the safety, tolerability and efficacy profiles of NOX-100 to reduce the number of intradialytic hypotension episodes. At single-blind stage I, the eligible subject will receive a 1-week run-in period followed by a 1-week NOX-100 treatment in a dose of 0.4mg/kg/hr. To evaluate the clearance of NOX-100, plasma levels of NOX-100 at the end of the 1st dialysis and prior to the 2nd dialysis will be measured. An interim analysis will be undertaken after the completion of first stage. The following process should be conducted only if the plasma level of NOX-100 decreases by 90% or more in these patients and all safety data have been reviewed by the medical monitor.

At double blind stage II, patients will be randomized to one of the following treatment sequences in a 1:1 ratio.

* Sequence A: NOX-100 treatment phase followed by Placebo treatment phase
* Sequence B: Placebo treatment phase followed by NOX-100 treatment phase

After a 1-week placebo, the subjects will receive the two 4-week treatment (sequence A or sequence B)which are separated by 1-week wash-out. In the NOX-100 treatment phase, subjects will subsequently receive NOX-100 in doses of 1.2, 2.5, 5, and 10 mg/kg/hr at the first three dialysis sessions over each week. In the placebo treatment phase, subjects will receive comparative placebo for four weeks. For the first 20 subjects, the treatment dose could be escalated only after the individual safety data have been reviewed by an unblinded medical monitor.

To confirm if there is hepatic metabolism of NOX-100 between dialysis sessions, a pre-dialysis plasma level will be tested at the 2nd dialysis of Week 2, 5, 7 and 10 in the second stage.

In both stages, the blood pressure will be measured pre-HD, every 30 minutes during HD and post-HD for monitoring the hypotension episode. For safety assessment, all AE(s), SAE(s) and any signs/symptoms during HD will be recorded. The safety of study drug will be followed until 4 weeks after last treatment.

A Data and Safety Monitoring Board (DSMB) will be established prior to start of the trial and the DSMB meeting will be hold every 6~12 months during study period. Both medical monitor and DSMB will be responsible for safeguarding the interests of trial participants.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-lactating females 20-80 years of age
* Patients who are hemodialysis dependent with a history of end-stage renal disease (ESRD) for at least 3 months and need at least three HD sessions per week
* History of intradialytic hypotension defined by at least 4 episodes with a fall in SBP of > 20 mmHg within 30 days prior to signing the ICF. At least two of the episodes must have caused symptoms requiring an intervention
* No change in anti-hypertensive regimen for at least one month prior to enrollment/randomization
* Be willing to sign the Informed Consent Form

Exclusion Criteria:

* Subjects with adequate laboratory results at screening
* Subjects with major psychiatric illness
* Subjects with history of arrhythmia or severe congestive heart failure (New York Heart Association (NYHA) Class III and IV) within past 6 months, or those with hypoxic myocardium confirmed by EKG
* Subjects with history of cirrhosis
* Subjects with active infection disease defined as current treatment with anti-infection agent(s)
* Subjects who need to receive nitrate and nitrite medication(s) (such as nitroglycerin, isosorbide mononitrate, and isosorbide dinitrate) for regular treatment
* Subjects who need to receive unstable dose of midodrine, etilefrine or amezinium treatment within 7 days prior to receive the study treatment.
* More than 14 drinks of alcohol per week
* Use of any investigational drug or participation in any drug study within 30 days prior to enrollment/randomization
* Any clinical condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk to participate in the study or confounds the ability to interpret data from the study as judged by the investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of hypotension episode requiring intervention | 10 weeks
  Number reduction of symptomatic hypotension requiring intervention during HD with NOX-100 treatment.

SECONDARY OUTCOMES:
systolic blood pressure (SBP) | 10 weeks
  Change in systolic blood pressure
Onset of symptoms of hypotension during HD | 10 weeks
  Time to onset of symptoms of hypotension during HD
The need for treatment intervention to raise BP. | 10 weeks
  Time to conduct a treatment intervention to raise BP

CONTACTS AND LOCATIONS:
Overall Officials: Monte Lai, Ph.D., Study Chair — Medinox, Inc.
Locations (6):
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Keelung Chang Gung Memorial Hospital, Keelung
  - Far Eastern Memorial Hospital, New Taipei City
  - Buddhist TzuChi General Hospital, Taipei Branch, New Taipei City
  - China Medical University Hospital, Taichung
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei